CLINICAL TRIAL: NCT01736553
Title: Spinal Muscular Atrophy (SMA) Biomarkers in the Immediate Postnatal Period of Development
Brief Title: Spinal Muscular Atrophy (SMA) Biomarkers Study in the Immediate Postnatal Period of Development
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Cure SMA (Other); Massachusetts General Hospital (Other); University of Iowa (Other)
Responsible Party: Principal Investigator, Stephen J. Kolb, Prinicipal Investigator of NeuroNEXT, Ohio State University
Other Study IDs: NN101; U01NS079163 (NIH)
Record Dates: First submitted 2012-11-19; First posted 2012-11-29 (Estimated); Results first posted 2018-05-04 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2018-04

CONDITIONS: Spinal Muscular Atrophy (SMA)
Keywords: Spinal Muscular Atrophy (SMA) Biomarkers; Healthy controls; Infants
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Absolute quantification of full length survival motor neuron (SMN) transcripts will be performed. The SMN1 and SMN2 transcripts will be measured in a multiplex reaction and SMN-del7 will be quantified separately. Droplet digital PCR will be used to determine SMN levels to further increase reliability and reduce variance in the SMN mRNA level determination. SMN protein in PBMCs SMN cell-based immunoassays will be performed. This assay is performed using a single monoclonal antibody for SMN and does not involve the disruption of cells. From the same PBMC sample, a commercially available SMN ELISA will also be performed according to the manufacturer's instructions. The B for SMA pilot study identified over 100 protein analytes that significantly correlated with motor function in SMA patients compared to controls.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Infants with Spinal Muscular Atrophy: Infants diagnosed Spinal Muscular Atrophy
- Healthy controls: Healthy control infants

SUMMARY:
Spinal muscular atrophy (SMA) is the leading genetic cause of death of infants. Strong preclinical evidence suggests that effective therapy must be delivered as early as possible to prevent progression of the disease. The primary study objective will be to identify prognostic and surrogate biomarkers of disease progression that will facilitate the execution of therapeutic SMA clinical trials in infants.

DETAILED DESCRIPTION:
Aim 1. To establish the validity of putative physiological SMA biomarkers in the immediate postnatal period. A longitudinal, natural history examination of physiological markers of muscle innervation will be performed in healthy and SMA infants. The first week of life is the ideal first time point, with visits occurring at scheduled visits up to the age two. Compound motor action potential (CMAP) amplitude and electrical impedance myography (EIM) will be examined and will be correlated with motor function. Each of these is associated with muscle innervation and provides information on the number and function of lower motor neurons in the spinal cord, the cellular target of SMA therapeutic interventions. This trial will establish the natural history of these putative SMA biomarkers as the disease evolves in affected infants. Moreover, our approach will allow for measurements in pre-symptomatic and early symptomatic subjects and determine their predictive value.

Aim 2. To establish the validity of putative molecular SMA biomarkers in the immediate postnatal period. Survival Motor Neuron (SMN2) copy number is a valid, predictive molecular SMA biomarker; however, it is fixed, and therefore not useful as a biomarker of clinical progression or response to therapy. SMN messenger Ribonucleic acid (mRNA) ( and protein expression is variable in different cell types and, in mice, naturally decreases with age postnatally. In this study, SMN expression levels will be measured longitudinally in SMA patients and controls. Additional putative molecular SMA markers that have been identified to correlate with motor function will be determined in an effort to distinguish between predictive markers that change prior to development of weakness and those that change as a consequence of weakness.

ELIGIBILITY:
Inclusion Criteria:

All infants will be between 0-6 months of age at the time of enrollment. Parents or guardians of the enrolled infants must sign an informed consent form prior to any study procedure being performed.

The infants with SMA must have already had a positive DNA test outside of the study to qualify for enrollment. An infant with SMA can have any number of SMN2 gene copies. Knowledge of the number of SMN2 gene copies prior to enrollment is not required.

Healthy control infants who meet the following criteria will be enrolled:

* Birth between 36 and 42 weeks inclusive of gestation
* Siblings of children with SMA must have had prior SMA genetic testing completed con-firming the infant is a healthy control
* Principal investigator feels the family/infant is able and willing to comply with study procedures
* Parent or guardian able to give informed consent

SMA infants who meet the following criteria will be enrolled:

* Birth between 36 and 42 weeks inclusive of gestation
* Positive SMN1 gene mutation/deletion
* Principal investigator feels the family/infant is able and willing to comply with study procedures
* Parent or guardian able to give informed consent

Exclusion Criteria:

* Use of any putative therapy intended to increase the amount of SMN protein in cells
* Enrollment in an SMA therapeutic trial at the time of enrollment in the SMA biomarker study
* Have a systemic illness requiring ongoing treatment, such as pneumonia
* Clinically significant abnormal findings (as determined by the investigator) on the physical examination or medical history (including history of tracheostomy tubes and ventilator-dependency)
* Dependency upon non-invasive ventilatory support (ie: BiPAP) for more than 12 hours/day

Max Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Fifty four (54) volunteers will be enrolled at 15 NeuroNEXT Network centers. Any volunteer who signs an informed consent form and has blood collected for the study is considered enrolled.
  Recruitment will be coordinated nationally through the Families of SMA Patient Network and NeuroNEXT who will help with the following:
  * Identifying infants diagnosed genetically with SMA because of a clinical suspicion prior to 6 months of age.
  * Publicize the project to raise awareness in medical and non-medical communities.
  Any normal infant may enroll in this study.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2012-12; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Kolb, MD PhD, Principal Investigator — Ohio State University
Locations (15):
- United States (15):
  - University of California - Davis, Davis, California
  - University of California - Los Angeles, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Mercy Hospital, Kansas City, Missouri
  - Washington University in St. Louis School of Medicine, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - State University of New York Upstate Medical Center, Syracuse, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - Doernbecher Children's Hospital, Portland, Oregon
  - Vanderbilt University, Nashville, Tennessee
  - Children's Medical Center of Dallas, Dallas, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah

REFERENCES:
- [Background] Campbell SK, Swanlund A, Smith E, Liao PJ, Zawacki L. Validity of the TIMPSI for estimating concurrent performance on the test of infant motor performance. Pediatr Phys Ther. 2008 Spring;20(1):3-10. doi: 10.1097/PEP.0b013e31815f66a6. PMID 18300928
- [Background] Dominguez E, Marais T, Chatauret N, Benkhelifa-Ziyyat S, Duque S, Ravassard P, Carcenac R, Astord S, Pereira de Moura A, Voit T, Barkats M. Intravenous scAAV9 delivery of a codon-optimized SMN1 sequence rescues SMA mice. Hum Mol Genet. 2011 Feb 15;20(4):681-93. doi: 10.1093/hmg/ddq514. Epub 2010 Nov 30. PMID 21118896
- [Background] Finkel RS, Hynan LS, Glanzman AM, Owens H, Nelson L, Cone SR, Campbell SK, Iannaccone ST; AmSMART Group. The test of infant motor performance: reliability in spinal muscular atrophy type I. Pediatr Phys Ther. 2008 Fall;20(3):242-6. doi: 10.1097/PEP.0b013e318181ae96. PMID 18703961
- [Background] Foust KD, Wang X, McGovern VL, Braun L, Bevan AK, Haidet AM, Le TT, Morales PR, Rich MM, Burghes AH, Kaspar BK. Rescue of the spinal muscular atrophy phenotype in a mouse model by early postnatal delivery of SMN. Nat Biotechnol. 2010 Mar;28(3):271-4. doi: 10.1038/nbt.1610. Epub 2010 Feb 28. PMID 20190738 (Retraction: PMID 36203015 Nat Biotechnol. 2022 Nov;40(11):1692)
- [Background] Hua Y, Sahashi K, Hung G, Rigo F, Passini MA, Bennett CF, Krainer AR. Antisense correction of SMN2 splicing in the CNS rescues necrosis in a type III SMA mouse model. Genes Dev. 2010 Aug 1;24(15):1634-44. doi: 10.1101/gad.1941310. Epub 2010 Jul 12. PMID 20624852
- [Background] Kolb SJ, Gubitz AK, Olszewski RF Jr, Ottinger E, Sumner CJ, Fischbeck KH, Dreyfuss G. A novel cell immunoassay to measure survival of motor neurons protein in blood cells. BMC Neurol. 2006 Feb 1;6:6. doi: 10.1186/1471-2377-6-6. PMID 16451734
- [Background] Kolb SJ, Kissel JT. Spinal muscular atrophy: a timely review. Arch Neurol. 2011 Aug;68(8):979-84. doi: 10.1001/archneurol.2011.74. Epub 2011 Apr 11. PMID 21482919
- [Background] Le TT, McGovern VL, Alwine IE, Wang X, Massoni-Laporte A, Rich MM, Burghes AH. Temporal requirement for high SMN expression in SMA mice. Hum Mol Genet. 2011 Sep 15;20(18):3578-91. doi: 10.1093/hmg/ddr275. Epub 2011 Jun 13. PMID 21672919
- [Background] Lutz CM, Kariya S, Patruni S, Osborne MA, Liu D, Henderson CE, Li DK, Pellizzoni L, Rojas J, Valenzuela DM, Murphy AJ, Winberg ML, Monani UR. Postsymptomatic restoration of SMN rescues the disease phenotype in a mouse model of severe spinal muscular atrophy. J Clin Invest. 2011 Aug;121(8):3029-41. doi: 10.1172/JCI57291. Epub 2011 Jul 25. PMID 21785219
- [Background] Morton JP, MacLaren DP, Cable NT, Bongers T, Griffiths RD, Campbell IT, Evans L, Kayani A, McArdle A, Drust B. Time course and differential responses of the major heat shock protein families in human skeletal muscle following acute nondamaging treadmill exercise. J Appl Physiol (1985). 2006 Jul;101(1):176-82. doi: 10.1152/japplphysiol.00046.2006. Epub 2006 Mar 24. PMID 16565353
- [Background] Narver HL, Kong L, Burnett BG, Choe DW, Bosch-Marce M, Taye AA, Eckhaus MA, Sumner CJ. Sustained improvement of spinal muscular atrophy mice treated with trichostatin A plus nutrition. Ann Neurol. 2008 Oct;64(4):465-70. doi: 10.1002/ana.21449. PMID 18661558
- [Background] Passini MA, Bu J, Richards AM, Kinnecom C, Sardi SP, Stanek LM, Hua Y, Rigo F, Matson J, Hung G, Kaye EM, Shihabuddin LS, Krainer AR, Bennett CF, Cheng SH. Antisense oligonucleotides delivered to the mouse CNS ameliorate symptoms of severe spinal muscular atrophy. Sci Transl Med. 2011 Mar 2;3(72):72ra18. doi: 10.1126/scitranslmed.3001777. PMID 21368223
- [Background] Piper MC, Pinnell LE, Darrah J, Maguire T, Byrne PJ. Construction and validation of the Alberta Infant Motor Scale (AIMS). Can J Public Health. 1992 Jul-Aug;83 Suppl 2:S46-50. PMID 1468050
- [Background] Porensky PN, Mitrpant C, McGovern VL, Bevan AK, Foust KD, Kaspar BK, Wilton SD, Burghes AH. A single administration of morpholino antisense oligomer rescues spinal muscular atrophy in mouse. Hum Mol Genet. 2012 Apr 1;21(7):1625-38. doi: 10.1093/hmg/ddr600. Epub 2011 Dec 20. PMID 22186025
- [Background] Rutkove SB, Shefner JM, Gregas M, Butler H, Caracciolo J, Lin C, Fogerson PM, Mongiovi P, Darras BT. Characterizing spinal muscular atrophy with electrical impedance myography. Muscle Nerve. 2010 Dec;42(6):915-21. doi: 10.1002/mus.21784. PMID 21104866
- [Background] Tiziano FD, Pinto AM, Fiori S, Lomastro R, Messina S, Bruno C, Pini A, Pane M, D'Amico A, Ghezzo A, Bertini E, Mercuri E, Neri G, Brahe C. SMN transcript levels in leukocytes of SMA patients determined by absolute real-time PCR. Eur J Hum Genet. 2010 Jan;18(1):52-8. doi: 10.1038/ejhg.2009.116. PMID 19603064
- [Background] Valori CF, Ning K, Wyles M, Mead RJ, Grierson AJ, Shaw PJ, Azzouz M. Systemic delivery of scAAV9 expressing SMN prolongs survival in a model of spinal muscular atrophy. Sci Transl Med. 2010 Jun 9;2(35):35ra42. doi: 10.1126/scitranslmed.3000830. PMID 20538619

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 12/2012 first subject enrolled, 9/2014 Enrollment Complete, 8/2015 Last Subject Visit
Pre-assignment Details: Subject's had staggered enrollment into the study based upon when identified with SMA. Participants could have visits at 0 and 3 months of age. We tried to enroll as early as possible, but only reported the data starting at 6months. 6 months was when the official visits began.
Period: Overall Study
Arm/Group | Infants With Spinal Muscular Atrophy | Healthy Controls
Started | 26 | 27
Completed | 7 | 23
Not Completed | 19 | 4
Not completed — Death | 12 | 0
Not completed — Withdrawal by Subject | 5 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Infants With Spinal Muscular Atrophy | Healthy Controls | Total
Number analyzed (Participants) | 26 | 27 | 53
Age, Continuous [Mean (Standard Deviation); unit: Weeks] — Gestational age at birth is reported.
  Weeks | 39 (1.5) | 39 (1.4) | 39 (1.45)
Age, Customized [Count of Participants; unit: Participants] — Age at Enrollment
  Participants
    Age at Enrollment: 0-2 Months | 4 | 10 | 14
    Age at Enrollment: 2-4 Months | 16 | 9 | 25
    Age at Enrollment: 5-6 Months | 6 | 8 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 11 | 13 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 3 | 9
  Not Hispanic or Latino | 20 | 24 | 44
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 1 | 2
  White | 24 | 21 | 45
  More than one race | 0 | 3 | 3
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26 | 27 | 53
SMN2 Copy Number [Count of Participants; unit: Participants]
  1 | 0 | 12 | 12
  2 | 16 | 13 | 29
  3 | 5 | 1 | 6
  4 | 1 | 0 | 1
  Unknown | 4 | 1 | 5
Birth Weight [Mean (Standard Deviation); unit: lbs] | 7 (1.2) | 7 (1.4) | 7 (1.3)
Birth Length [Mean (Standard Deviation); unit: inches] | 20 (1.2) | 20 (1.0) | 20 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Motor Function Assessments- Test for Infant Motor Performance Screening Items (TIMPSI)
Description: Describe & compare the distribution of motor function assessments over the first two years of life in SMA vs. healthy control infants.
  The TIMPSI is used to assess the postural and selective control of movement typically used by infants younger than 5 months. The TIMPSI scores were related to an infant's ability to reach. The TIMPSI is a 29-item evaluation that contains 3 item sets: a Screening set, an Easy set, and a Hard set. The Screening set consists of 11 items from the TIMP, each with a 5- to 7-point rating scale; the Easy set has 6 items with 5- or 6-point rating scales and 4 dichotomously scored items; the Hard set has 8 items, 3 with 5-point rating scales and 5 items that are scored dichotomously. The Total score is derived from all subset scores and is the sum of those subset scores. The final score could range from 0 to 99 points. The higher the score the better the functional ability of the participant. Linear mixed effects models were used for analyses.
Time Frame: Up to 24 months
Population: The overall number of participants analyzed (19 and 26) differs from the total enrollment in each cohort reported in the participant flow (26 and 27, respectively) because of the staggered enrollment and significant mortality.
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Infants With Spinal Muscular Atrophy | Healthy Controls
Number analyzed (Participants) | 19 | 26
scores on a scale
  6 month | 36.06 [27.20 to 44.91] | 88.47 [80.52 to 96.43]
  9 month: number analyzed (Participants) | 11 | 26
  9 month | 40.54 [29.91 to 51.18] | 89.44 [81.47 to 97.41]
  12 month: number analyzed (Participants) | 12 | 26
  12 month | 32.03 [21.39 to 42.68] | 85.39 [77.41 to 93.36]
  18 month: number analyzed (Participants) | 4 | 23
  18 month | 26.35 [10.87 to 41.83] | 87.35 [79.12 to 95.57]
  24 month: number analyzed (Participants) | 7 | 21
  24 month | 23.14 [10.04 to 36.23] | 88.65 [80.19 to 97.11]

2. Primary Outcome: Motor Function Assessments- The Children's Hospital of Philadelphia Infant Test for Neuromuscular Disorders (CHOP-INTEND)
Description: The TIMPSI motor function testing was done during all of the study visits knowing that the healthy controls would eventually ceiling out. The study design allowed for secondary motor function tests based on the score of the TIMPSI. If infants scored a 41 or above on the TIMPSI they would be tested with the AIMS. If they were below they were tested with the CHOP-INTEND. The CHOP-INTEND is a reliable and validated, comprehensive assessment of the postural and selective control of movement needed by infants. It is a clinician-rated questionnaire developed to assess motor skill in spinal muscular atrophy type I. The 16 items are scored from 0 to 4. The global score ranges from 0 to 64, a higher score indicating better motor skills.(Finkel, McDermott, 2014). All healthy controls based upon scores at 6 months moved on to the AIMS test, therefore no healthy controls completed the CHOP-INTEND. Linear mixed effects models were used for analyses of Motor function outcome data.
Time Frame: Up to 24 months
Population: Patients enrolled in the trial from birth. The overall number of participants analyzed (14 and 0) differs from the total enrollment in each cohort reported in the participant flow (26 and 27, respectively) because of the staggered enrollment, significant mortality, and protocol design of who was eligible for this second motor measure.
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Infants With Spinal Muscular Atrophy
Number analyzed (Participants) | 14
scores on a scale
  6 month | 18.38 [15.02 to 21.75]
  9 month: number analyzed (Participants) | 6
  9 month | 13.18 [9.24 to 17.12]
  12 month: number analyzed (Participants) | 7
  12 month | 9.74 [5.01 to 14.46]
  18 month: number analyzed (Participants) | 2
  18 month | 7.52 [2.89 to 12.16]
  24 month: number analyzed (Participants) | 3
  24 month | 7.01 [6.82 to 7.19]

3. Primary Outcome: Motor Function Assessments-Alberta Infant Motor Scale (AIMS)
Description: Linear mixed effects models were used for analyses.
  The reason that the number of infants differ from those in participant flow is based upon the protocol. The selection of which secondary test to perform depended upon the score of the TIMPSI that was performed. TIMPSI <41, do CHOP-NTEND. TIMPSI > 41, do AIMS.
  The AIMS incorporates the neuromaturational concept and the dynamical systems theory and is used to measure gross motor maturation of infants from birth through the age of independent walking (Piper, Pinnell et al. 1992, Piper, Darrah et al 1994). In the AIMS, the impact of neurological components on motor development is reflected by a sequence of motor skills, which are used as the basis of assessment. The AIMS consists of 58 items, including 4 positions: prone (21 items), supine (9 items), sitting (12 items) & standing(16 items). The highest score available is 58. The higher the score the better the functional ability of the participant.
Time Frame: Up to 24 months
Population: Patients enrolled in the trial from birth to 6 months of age. The overall number of participants analyzed (5 and 26) differs from the total enrollment in each cohort reported in the participant flow (26 and 27) because of the staggered enrollment, significant mortality and protocol design of who was eligible for this second motor measure.
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Infants With Spinal Muscular Atrophy | Healthy Controls
Number analyzed (Participants) | 5 | 26
Scores on a scale
  6 month: number analyzed (Participants) | 5 | 25
  6 month | 11.74 [3.91 to 19.58] | 19.29 [16.4 to 22.19]
  9 month: number analyzed (Participants) | 4 | 26
  9 month | 15.58 [2.51 to 28.64] | 34.10 [29.05 to 39.14]
  12 month: number analyzed (Participants) | 5 | 25
  12 month | 21.60 [6.66 to 36.53] | 37.10 [30.52 to 43.68]
  18 month: number analyzed (Participants) | 3 | 24
  18 month | 19.18 [2.03 to 36.32] | 38.62 [31.30 to 45.93]
  24 month: number analyzed (Participants) | 4 | 22
  24 month | 14.71 [2.17 to 27.25] | 37.76 [29.81 to 45.71]

4. Primary Outcome: Putative Physiological Biomarker- Compound Motor Action Potential Testing (CMAP)
Description: Describe and compare the distribution of the putative physiological and molecular biomarkers over the first two years of life in SMA vs. healthy control infants.
  Maximum ulnar CMAP amplitude and area will be obtained by recording from the abductor digitiminimi muscle following ulnar nerve stimulation at the wrist. All electrophysiologic testing will be performed by certified electromyographers experienced in the assessment of pediatric patients. Maximum values for both negative peak (NP) amplitude and NP area will be obtained. No medications will be used.
  This test is done routinely in this population. Pediatric electrodes and each site's standard electromyograph devices will be utilized. The test, while not considered to be painful, may cause some discomfort similar to a static electric shock. Infants may whimper or cry due to the surprise of the shock. Each shock lasts approximately 0.1 millisecond. The testing duration is expected to be approximately 30 seconds.
Time Frame: Up to 24 months
Population: Patients enrolled in the trial from birth to 6 months. The overall number of participants analyzed (18/ and 26) differs from the total enrollment in the participant flow (26 and 27) because of the staggered enrollment, significant mortality and tolerance of procedure. Therefore not all infants enrolled were included in all longitudinal analyses.
Measure: Mean (95% Confidence Interval); unit: mV
Arm/Group | Infants With Spinal Muscular Atrophy | Healthy Controls
Number analyzed (Participants) | 18 | 26
mV
  6 month | 1.07 [0.17 to 1.96] | 6.00 [5.22 to 6.78]
  12 month: number analyzed (Participants) | 11 | 25
  12 month | 0.51 [-0.56 to 1.59] | 5.95 [5.16 to 6.75]
  18 month: number analyzed (Participants) | 5 | 24
  18 month | 0.49 [-0.98 to 1.95] | 6.55 [5.75 to 7.36]
  24 month: number analyzed (Participants) | 6 | 21
  24 month | -0.02 [-1.46 to 1.42] | 6.74 [5.91 to 7.58]

5. Primary Outcome: Molecular Biomarkers- mRNA
Description: Describe and compare the distribution of the putative physiological and molecular biomarkers over the first two years of life in SMA vs. healthy control infants.
  Results were measured in survival motor neurons (SMN), hypoxanthine phosphoribosyltransferase (HPRT) Ratio.
Time Frame: Up to 24 months
Population: Patients enrolled in the trial from birth to 6 months. The overall number of participants analyzed (19 and 22) differs from the total enrollment in the participant flow (26 and 27) because of the staggered enrollment, significant mortality, & insufficient sample. Therefore not all infants enrolled were included in all longitudinal analyses.
Measure: Mean (95% Confidence Interval); unit: SMN/HPRT Ratio
Arm/Group | Infants With Spinal Muscular Atrophy | Healthy Controls
Number analyzed (Participants) | 19 | 22
SMN/HPRT Ratio
  6 month | 0.55 [0.39 to 0.71] | 1.29 [1.14 to 1.44]
  12 month: number analyzed (Participants) | 10 | 21
  12 month | 0.47 [0.26 to 0.69] | 1.21 [1.06 to 1.37]
  18 month: number analyzed (Participants) | 5 | 22
  18 month | 0.50 [0.19 to 0.80] | 1.11 [0.96 to 1.26]
  24 month: number analyzed (Participants) | 5 | 17
  24 month | 0.66 [0.35 to 0.97] | 1.20 [1.03 to 1.37]

6. Primary Outcome: Molecular Biomarkers- SMN Protein Levels
Description: Describe and compare the distribution of the putative physiological and molecular biomarkers over the first two years of life in SMA vs. healthy control infants.
Time Frame: Up to 24 months
Population: Patients enrolled in the trial from birth to 6 months. The overall number of participants analyzed (15 and 18) differs from the total enrollment reported in the participant flow (26 and 27) because of the staggered enrollment, significant mortality, insufficient sample. Therefore not all infants enrolled were included in all longitudinal analyses.
Measure: Mean (95% Confidence Interval); unit: pg/10^7 PBMC
Arm/Group | Infants With Spinal Muscular Atrophy | Healthy Controls
Number analyzed (Participants) | 15 | 18
pg/10^7 PBMC
  6 month | 4798.85 [2799.07 to 6798.63] | 8325.96 [6435.08 to 10217]
  12 month: number analyzed (Participants) | 8 | 17
  12 month | 6719.63 [4404.92 to 9034.3] | 10247 [8228.29 to 12265]
  18 month: number analyzed (Participants) | 5 | 14
  18 month | 3108.79 [476.39 to 5741.19] | 6635.90 [4401.46 to 8870.34]
  24 month: number analyzed (Participants) | 3 | 12
  24 month | 8502.48 [5562.01 to 11443] | 12030 [9552.13 to 14507]

7. Primary Outcome: Putative Physiological Biomarkers-Weight
Description: as for outcome 6
Time Frame: Up to 24 months
Population: Subjects enrolled from birth to 6 months. The overall number of participants analyzed (19 and 26) differs from the total enrollment reported in the participant flow (26 and 27) because of the staggered enrollment & significant mortality. Therefore not all infants enrolled were included in all longitudinal analyses.
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Infants With Spinal Muscular Atrophy | Healthy Controls
Number analyzed (Participants) | 19 | 26
kg
  6 month: number analyzed (Participants) | 19 | 25
  6 month | 6.88 [6.46 to 7.31] | 7.83 [7.43 to 8.23]
  9 month: number analyzed (Participants) | 11 | 26
  9 month | 7.92 [7.34 to 8.49] | 8.94 [8.51 to 9.37]
  12 month: number analyzed (Participants) | 12 | 26
  12 month | 8.71 [8.10 to 9.33] | 9.88 [9.41 to 10.36]
  18 month: number analyzed (Participants) | 5 | 24
  18 month | 9.95 [9.17 to 10.72] | 11.40 [10.95 to 11.85]
  24 month: number analyzed (Participants) | 7 | 22
  24 month | 10.47 [9.71 to 11.23] | 12.74 [12.25 to 13.23]

8. Primary Outcome: Correlation of Biomarkers With Motor Function Tests for SMA Subjects- CMAP
Description: In these analyses motor function score was the outcome measure. Correlation was defined as the estimated mean increase per a one unit increase in the biomarker under consideration. A linear mixed effects model was used to estimate the correlation between the biomarker and motor function score. Separate models were used for the TIMPSI and CHOP-INTEND. In the CHOP-INTEND analyses, correlations were not estimable for the 18 and 24 month visits.
Time Frame: up to 24 months
Population: The overall number of participants analyzed (19 and 14) differs from the total enrollment reported in the participant flow (26) because of the staggered enrollment and significant mortality. Therefore not all infants enrolled were included in all longitudinal analyses.
Measure: Mean (95% Confidence Interval); unit: mV/scale unit
Arm/Group | Correlation With TIMPSI | Correlation With CHOP-INTEND
Number analyzed (Participants) | 19 | 14
mV/scale unit
  6 month | 9.36 [5.59 to 13.13] | 17.25 [-2.26 to 36.77]
  12 month: number analyzed (Participants) | 12 | 7
  12 month | 22.88 [16.24 to 29.52] | 21.53 [-34.94 to 78.00]
  18 month: number analyzed (Participants) | 4 | 0
  18 month | 17.48 [9.07 to 25.89] |
  24 month: number analyzed (Participants) | 7 | 0
  24 month | 18.57 [10.03 to 27.11] |

9. Primary Outcome: Correlation of Biomarkers With Motor Function Tests for SMA Subjects- mRNA
Description: In these analyses motor function score was the outcome measure. Correlation was defined as the estimated mean increase per a one unit increase in the biomarker under consideration. A linear mixed effects model was used to estimate the correlation between the biomarker and motor function score. Separate models were used for the TIMPSI and CHOP-INTEND.
Time Frame: up to 24 months
Measure: Mean (95% Confidence Interval); unit: (SMN/HPRT ratio)/scale unit
Arm/Group | Correlation With TIMPSI | Correlation With CHOP-INTEND
Number analyzed (Participants) | 26 | 26
(SMN/HPRT ratio)/scale unit
  6 month | 53.60 [-0.04 to 107.24] | 0.11 [-15.81 to 16.03]
  12 month | 125.52 [40.81 to 210.22] | 0.11 [-15.81 to 16.03]
  18 month | 181.22 [3.65 to 358.78] | 0.11 [-15.81 to 16.03]
  24 month | 46.43 [-12.65 to 105.51] | 0.11 [-15.81 to 16.03]

10. Primary Outcome: Correlation of Biomarkers With Motor Function Tests for SMA Subjects- SMN Protein
Description: In these analyses motor function score was the outcome measure. Correlation was defined as the estimated mean increase per a one unit increase in the biomarker under consideration. A linear mixed effects model was used to estimate the correlation between the biomarker and motor function score. Separate models were used for the TIMPSI and CHOP-INTEND. In the CHOP-INTEND analyses, the correlation at the 24 month visit was not estimable.
Time Frame: up to 24 months
Population: The overall number of participants analyzed (14 and 19) differs from the total enrollment reported in the participant flow (26) because of the staggered enrollment and significant mortality. Therefore not all infants enrolled were included in all longitudinal analyses.
Measure: Mean (95% Confidence Interval); unit: (pg/10^7 PBMC)/scale unit
Arm/Group | Correlation With CHOP-INTEND | Correlation With TIMPSI
Number analyzed (Participants) | 14 | 19
(pg/10^7 PBMC)/scale unit
  6 month | -0.0011 [-0.0053 to 0.0032] | -0.0003 [-0.0033 to 0.0027]
  12 month: number analyzed (Participants) | 7 | 12
  12 month | 0.00066 [-0.0057 to 0.0071] | -0.0003 [-0.00033 to 0.0027]
  18 month: number analyzed (Participants) | 2 | 4
  18 month | 0.026 [-0.0093 to 0.061] | -0.0003 [-0.00033 to 0.0027]
  24 month: number analyzed (Participants) | 0 | 7
  24 month |  | -0.0003 [-0.00033 to 0.0027]

11. Primary Outcome: Correlation of Biomarkers With Motor Function Tests for SMA Subjects- Weight
Description: as for outcome 9
Time Frame: up to 24 months
Measure: Mean (95% Confidence Interval); unit: kg/scale unit
Arm/Group | Correlation With TIMPSI | Correlation With CHOP-INTEND
Number analyzed (Participants) | 26 | 26
kg/scale unit | 2.27 [-3.34 to 7.87] | -2.39 [-4.13 to -0.65]

12. Primary Outcome: Correlation of Biomarkers With Motor Function Tests for Healthy Control Subjects- CMAP
Description: In these analyses motor function score was the outcome measure. Correlation was defined as the estimated mean increase per a one unit increase in the biomarker under consideration. A linear mixed effects model was used to estimate the correlation between the biomarker and motor function score. Separate models were used for the TIMPSI and AIMS.
Time Frame: up to 24 months
Population: The overall number of participants analyzed (26 and 26) differs from the total enrollment reported in the participant flow at each visit (27) because of the staggered enrollment, significant mortality and tolerance of testing.
Measure: Mean (95% Confidence Interval); unit: mV/scale unit
Groups:
- Correlation With TIMPSI: Healthy Control Subjects Motor Test- TIMPSI correlated with the CMAP exam
- Correlation With AIMS: Healthy Control Subjects Motor Test- AIMS correlated with the CMAP exam
Arm/Group | Correlation With TIMPSI | Correlation With AIMS
Number analyzed (Participants) | 26 | 26
mV/scale unit
  6 month: number analyzed (Participants) | 26 | 25
  6 month | -0.23 [-2.88 to 2.43] | 0.21 [-0.63 to 1.05]
  12 month: number analyzed (Participants) | 26 | 25
  12 month | -4.52 [-7.53 to -1.51] | 0.21 [-0.63 to 1.05]
  18 month: number analyzed (Participants) | 23 | 24
  18 month | -0.58 [-3.07 to 1.92] | 0.21 [-0.63 to 1.05]
  24 month: number analyzed (Participants) | 21 | 22
  24 month | 1.14 [-2.05 to 4.34] | 0.21 [-0.63 to 1.05]

13. Primary Outcome: Correlation of Biomarkers With Motor Function Tests for Healthy Control Subjects- mRNA
Description: as for outcome 12
Time Frame: up to 24 months
Population: Labs were not obtainable for all subjects. The overall number of participants analyzed (26 and 26) differs from the total enrollment reported in the participant flow (27) because of the staggered enrollment, significant mortality and protocol design.
Measure: Mean (95% Confidence Interval); unit: (SMN/HPRT Ratio)/scale unit
Groups:
- Correlation With TIMPSI: Healthy Control Subjects Motor Test- TIMPSI correlated with the mRNA
- Correlation With AIMS: Healthy Control Subjects Motor Test- AIMS correlated with the mRNA
Arm/Group | Correlation With TIMPSI | Correlation With AIMS
Number analyzed (Participants) | 26 | 26
(SMN/HPRT Ratio)/scale unit | 9.52 [3.18 to 15.86] | -2.46 [-6.20 to 1.28]

14. Primary Outcome: Correlation of Biomarkers With Motor Function Tests for Healthy Control Subjects- Weight
Description: as for outcome 12
Time Frame: up to 24 months
Population: The overall number of participants analyzed (26 and 26) differs from the total enrollment reported in the participant flow (27) because of the staggered enrollment and significant mortality.
Measure: Mean (95% Confidence Interval); unit: kg/scale unit
Groups:
- Correlation With TIMPSI: Healthy Control Subjects Motor Test- TIMPSI correlated with weight
- Correlation With AIMS: Healthy Control Subjects Motor Test- AIMS correlated with weight
Arm/Group | Correlation With TIMPSI | Correlation With AIMS
Number analyzed (Participants) | 26 | 26
kg/scale unit
  6 month | 0.60 [-1.71 to 2.90] | 1.48 [-0.68 to 3.66]
  9 month | 0.60 [-1.71 to 2.90] | -0.72 [-4.06 to 2.62]
  12 month | 0.60 [-1.71 to 2.90] | 1.14 [-2.12 to 4.39]
  18 month | 0.60 [-1.71 to 2.90] | -0.46 [-4.39 to 3.47]
  24 month | 0.60 [-1.71 to 2.90] | 3.53 [-0.76 to 7.82]

15. Secondary Outcome: Biomarker Prediction of Risk of Death
Description: Examine whether any of the motor function assessments, putative physiological, or molecular biomarkers predict risk of death in the SMA cohort. Proportional hazards regression models used to determine if motor function scores, mRNA, and protein levels predict death in SMA subjects. Considered each predictor separately modeled as a time-varying covariate (predictor values were allowed to vary as time to death was assessed).
Time Frame: Up to 24 months
Measure: Mean (95% Confidence Interval); unit: Hazard Ratio
Groups:
- Estimated Hazard Ratio: Proportional hazards regression models used to determine if motor function scores, mRNA, and protein levels predict death in SMA subjects
Arm/Group | Estimated Hazard Ratio
Number analyzed (Participants) | 26
Hazard Ratio
  TIMPSI (per 10 unit increase) | 0.72 [0.50 to 1.04]
  CHOP-INTEND (per 10 unit increase) | 0.94 [0.59 to 1.51]
  CMAP Peak Amplitude (per 1 unit increase) | 0.37 [0.10 to 1.29]
  mRNA (per 1 unit increase) | 0.28 [0.0009 to 8.82]
  Protein Level (per 1000 unit increase) | 1.27 [0.98 to 1.65]
  Weight (per 10kg increase) | 0.02 [0.0004 to 1.28]

16. Secondary Outcome: Motor Function Assessments- Test for Infant Motor Performance Screening Items (TIMPSI) SMN Copy Number =2 Cohort
Description: Describe and compare the distribution of motor function assessments over the first two years of life in SMA subjects with SMN copy number = 2 versus healthy control infants.
  The TIMPSI is used to assess the postural and selective control of movement typically used by infants younger than 5 months. The TIMPSI scores were related to an infant's ability to reach. The TIMPSI is a 29-item evaluation that contains 3 item sets: a Screening set, an Easy set, and a Hard set. The Screening set consists of 11 items from the TIMP, each with a 5- to 7-point rating scale; the Easy set has 6 items with 5- or 6-point rating scales and 4 dichotomously scored items; the Hard set has 8 items, 3 with 5-point rating scales and 5 items that are scored dichotomously. The Total score is derived from all subset scores and is the sum of those subset scores. The final score could range from 0 to 99 points. The higher the score the better the functional ability of the participant.
Time Frame: Up to 24 months
Population: The overall number of participants analyzed (14 and 26) differs from the total enrollment reported in the participant flow (26 and 27 respectively) because of the staggered enrollment, subset of infants with SMN2 & significant mortality.
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Groups:
- Infants With Spinal Muscular Atrophy (SMN=2): Infants diagnosed Spinal Muscular Atrophy (SMN=2)
Arm/Group | Infants With Spinal Muscular Atrophy (SMN=2) | Healthy Controls
Number analyzed (Participants) | 14 | 26
Scores on a scale
  6 month | 24.53 [17.89 to 31.17] | 88.25 [83.34 to 93.15]
  9 month: number analyzed (Participants) | 6 | 26
  9 month | 20.08 [10.11 to 30.05] | 89.20 [84.29 to 94.11]
  12 month: number analyzed (Participants) | 7 | 26
  12 month | 13.82 [4.40 to 23.24] | 85.15 [80.24 to 90.06]
  18 month: number analyzed (Participants) | 2 | 23
  18 month | 8.82 [-8.24 to 25.89] | 87.36 [82.16 to 92.56]
  24 month: number analyzed (Participants) | 3 | 21
  24 month | 7.51 [-6.83 to 22.03] | 88.92 [83.49 to 94.36]

17. Secondary Outcome: Motor Function Assessments- The Children's Hospital of Philadelphia Infant Test for Neuromuscular Disorders (CHOP-INTEND) SMN Copy Number =2 Cohort
Description: Describe and compare the distribution of motor function assessments over the first two years of life in SMA subjects with SMN copy number = 2 versus healthy control infants.
  The CHOP-INTEND is a reliable and validated, comprehensive assessment of the postural and selective control of movement needed by infants. It is a clinician-rated questionnaire developed to assess motor skill in spinal muscular atrophy type I. The 16 items are scored from 0 to 4. The global score ranges from 0 to 64, a higher score indicating better motor skills.(Finkel, McDermott, 2014).
Time Frame: Up to 24 months
Population: The overall number of participants analyzed (14) differs from the total enrollment reported in the participant flow (26) because of the staggered enrollment, subset of infants with SMN2 , and significant mortality. Healthy controls did not complete this visit due to the protocol.
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Infants With Spinal Muscular Atrophy (SMN=2)
Number analyzed (Participants) | 14
Scores on a scale
  6 month | 18.05 [14.86 to 21.25]
  9 month: number analyzed (Participants) | 6
  9 month | 12.87 [8.93 to 16.81]
  12 month: number analyzed (Participants) | 7
  12 month | 9.38 [4.61 to 14.12]
  18 month: number analyzed (Participants) | 2
  18 month | 7.33 [2.39 to 12.26]
  24 month: number analyzed (Participants) | 3
  24 month | 7.00 [6.72 to 7.28]

18. Secondary Outcome: Putative Physiological Biomarker- Compound Motor Action Potential Testing (CMAP) SMN Copy Number = 2 Cohort
Description: Describe and compare the distribution of the putative physiological and molecular biomarkers over the first two years of life in SMA2 vs. healthy control infants.
  Maximum ulnar CMAP amplitude and area will be obtained by recording from the abductor digitiminimi muscle following ulnar nerve stimulation at the wrist. All electrophysiologic testing will be performed by certified electromyographers experienced in the assessment of pediatric patients. Maximum values for both negative peak (NP) amplitude and NP area will be obtained. No medications will be used.
  This test is done routinely in this population. Pediatric electrodes and each site's standard electromyograph devices will be utilized. The test, while not considered to be painful, may cause some discomfort similar to a static electric shock. Infants may whimper or cry due to the surprise of the shock. Each shock lasts approximately 0.1 millisecond. The testing duration is expected to be approximately 30 seconds.
Time Frame: Up to 24 months
Population: The overall number of participants analyzed (13 and 26) differs from the total enrollment in the participant flow (26 and 27) because of the staggered enrollment, subset of patients with SMA, significant mortality, and tolerance of procedure.
Measure: Mean (95% Confidence Interval); unit: mV
Arm/Group | Infants With Spinal Muscular Atrophy (SMN=2) | Healthy Controls
Number analyzed (Participants) | 13 | 26
mV
  6 month | 0.36 [-0.04 to 1.84] | 5.95 [5.30 to 6.60]
  12 month: number analyzed (Participants) | 7 | 25
  12 month | 0.33 [-0.54 to 1.19] | 5.92 [5.25 to 6.58]
  18 month: number analyzed (Participants) | 2 | 24
  18 month | 0.90 [-0.04 to 1.84] | 6.49 [5.80 to 7.19]
  24 month: number analyzed (Participants) | 0 | 21
  24 month |  | 6.63 [5.92 to 7.36]

19. Secondary Outcome: Molecular Biomarkers- mRNA SMA Copy Number = 2 Cohort
Description: as for outcome 6
Time Frame: Up to 24 months
Population: The overall number of participants analyzed (14 and 22) differs from the total enrollment in the participant flow (26 and 27) because of the staggered enrollment, subset of patients with SMA, significant mortality, and insufficient sample.
Measure: Mean (95% Confidence Interval); unit: SMN/HPRT Ratio
Arm/Group | Infants With Spinal Muscular Atrophy (SMN=2) | Healthy Controls
Number analyzed (Participants) | 14 | 22
SMN/HPRT Ratio
  6 month | 0.46 [0.31 to 0.62] | 1.29 [1.16 to 1.43]
  12 month: number analyzed (Participants) | 6 | 21
  12 month | 0.38 [0.31 to 0.45] | 1.21 [1.07 to 1.35]
  18 month: number analyzed (Participants) | 2 | 22
  18 month | 0.29 [0.08 to 0.49] | 1.12 [0.97 to 1.26]
  24 month: number analyzed (Participants) | 3 | 22
  24 month | 0.40 [0.19 to 0.61] | 1.23 [1.07 to 1.39]

20. Secondary Outcome: Molecular Biomarkers- SMN Protein Levels SMA Copy Number = 2
Description: Describe and compare the distribution of the putative physiological and molecular biomarkers over the first two years of life in SMA2 vs. healthy control infants.
Time Frame: Up to 24 months
Population: Patients enrolled in the trial at birth. The overall number of participants analyzed (10 and 18) differs from the total enrollment reported in the participant flow (26 and 27) because of the staggered enrollment, significant mortality, subset of SMA subjects, and insufficient sample.
Measure: Mean (95% Confidence Interval); unit: pg/10^7 PBMC
Arm/Group | Infants With Spinal Muscular Atrophy (SMN=2) | Healthy Controls
Number analyzed (Participants) | 10 | 18
pg/10^7 PBMC
  6 month | 3785.02 [1245.92 to 6324.12] | 8598.73 [6472.81 to 10725]
  12 month: number analyzed (Participants) | 4 | 17
  12 month | 5800.63 [2828.39 to 8772.87] | 10614 [8341.73 to 12887]
  18 month: number analyzed (Participants) | 2 | 14
  18 month | 1612.35 [-1753.19 to 4977.90] | 6426.06 [3892.03 to 8960.09]
  24 month: number analyzed (Participants) | 1 | 12
  24 month | 6912.88 [3225.48 to 10600] | 11727 [8930.09 to 14523]

21. Secondary Outcome: Putative Physiological Biomarkers-Weight SMN Copy Number =2 Cohort
Description: Describe and compare the distribution of motor function assessments over the first two years of life in SMA subjects with SMN copy number = 2 versus healthy control infants
Time Frame: Up to 24 months
Population: The overall number of participants analyzed (14 and 26) differs from the total enrollment reported in the participant flow (26 and 27) because of the staggered enrollment, subset of SMA subjects, and significant mortality. Therefore not all infants enrolled were included in all longitudinal analyses.
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Infants With Spinal Muscular Atrophy (SMN=2) | Healthy Controls
Number analyzed (Participants) | 14 | 26
kg
  6 month: number analyzed (Participants) | 14 | 25
  6 month | 6.63 [6.14 to 7.13] | 7.83 [7.43 to 8.23]
  9 month: number analyzed (Participants) | 6 | 26
  9 month | 7.70 [7.00 to 8.39] | 8.93 [8.50 to 9.36]
  12 month: number analyzed (Participants) | 7 | 26
  12 month | 8.51 [7.70 to 9.32] | 9.88 [9.40 to 10.37]
  18 month: number analyzed (Participants) | 2 | 24
  18 month | 9.65 [8.47 to 10.84] | 11.40 [10.93 to 11.87]
  24 month: number analyzed (Participants) | 3 | 22
  24 month | 9.77 [8.57 to 10.98] | 12.72 [12.23 to 13.22]

22. Secondary Outcome: Correlation of CMAP Biomarker With Motor Function Tests for SMA Subjects SMN Copy Number =2 Cohort
Description: Examine the correlation between each of the putative physiological and molecular biomarkers with the TIMPSI and CHOP-INTEND over the first two years of life in SMA (SMN = 2). All estimated correlations are the same at each study visit.
Time Frame: up to 24 months
Population: The overall number of participants with SMA analyzed (14/14) differs from the total enrollment reported in the participant flow (26) because of the staggered enrollment, subset of subjects with SMA and significant mortality.
Measure: Mean (95% Confidence Interval); unit: mV/scores on a scale
Groups:
- Correlation With TIMPSI; Correlation With CHOP-INTEND: Infants Diagnosed with SMN=2
Arm/Group | Correlation With TIMPSI | Correlation With CHOP-INTEND
Number analyzed (Participants) | 14 | 14
mV/scores on a scale | 5.10 [0.095 to 10.11] | 3.71 [-0.21 to 7.62]

23. Secondary Outcome: Correlation of mRNA Biomarkers With Motor Function Tests for SMA Subjects SMN Copy Number =2 Cohort
Description: as for outcome 22
Time Frame: up to 24 months
Population: The overall number of participants with SMA analyzed (14 and 14) differs from the total enrollment reported in the participant flow (26) because of the staggered enrollment, subset of subjects with SMA and significant mortality.
Measure: Mean (95% Confidence Interval); unit: (SMN/HPRT)/scores on a scale
Groups:
- Correlation With TIMPSI; Correlation With CHOP-INTEND: Infants diagnosed Spinal Muscular Atrophy (SMN=2)
Arm/Group | Correlation With TIMPSI | Correlation With CHOP-INTEND
Number analyzed (Participants) | 14 | 14
(SMN/HPRT)/scores on a scale | -6.39 [-28.59 to 15.80] | 0.097 [-16.08 to 16.27]

24. Secondary Outcome: Correlation of Protein Level Biomarkers With Motor Function Tests for SMA Subjects SMN Copy Number =2 Cohort
Description: as for outcome 22
Time Frame: up to 24 months
Population: The overall number of participants with SMA analyzed (10/10) differs from the total enrollment reported in the participant flow (26) because of the staggered enrollment, insufficient sample, subset of subjects with SMA and significant mortality.
Measure: Mean (95% Confidence Interval); unit: (pg/10^7 PBMC0/scores on a scale
Groups:
- Correlation With TIMPSI; Correlation With CHOP-INTEND: Infants diagnosed with SMA (SMN=2)
Arm/Group | Correlation With TIMPSI | Correlation With CHOP-INTEND
Number analyzed (Participants) | 10 | 10
(pg/10^7 PBMC0/scores on a scale | 0.000063 [-0.0012 to 0.0013] | 0.00048 [-0.00077 to 0.0017]

25. Secondary Outcome: Correlation of Biomarkers (Weight) With Motor Function Tests for SMA Subjects SMN Copy Number =2 Cohort
Description: as for outcome 22
Time Frame: up to 24 months
Population: as for outcome 22
Measure: Mean (95% Confidence Interval); unit: kg/scores on a scale
Arm/Group | Correlation With TIMPSI | Correlation With CHOP-INTEND
Number analyzed (Participants) | 14 | 14
kg/scores on a scale | -2.50 [-4.78 to -.23] | -2.43 [-4.19 to -0.67]

ADVERSE EVENTS:
Description: Since this trial was not a treatment study, Adverse Events (AEs) were only collected if they related to the procedures done at the visit. There were no AEs to report.
Arm/Group | Infants With Spinal Muscular Atrophy | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 12/26 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/27
Other Adverse Events (participants affected / at risk) | 0/26 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No